CLINICAL TRIAL: NCT05369884
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of WPQW Granule for Overlap of Non-Erosive Reflux Disease(NERD) and Diarrhea Predominant Diarrhea Irritable Bowel Syndrome(IBS-D)
Brief Title: Efficacy and Safety of WPQW Granule for Overlap of NERD and IBS-D
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Tianjin Nankai Hospital (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Shanxi University of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Yunnan Provinical Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYYCXTD-C-202010
Record Dates: First submitted 2022-05-08; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-12

CONDITIONS: Non-erosive Reflux Disease; Diarrhea-Predominant Irritable Bowel Syndrome
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators were masked to group assignment. An independent statistician was masked for the data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral administration of WPQW granule with warm water，2 sachets each time, 3 times a day, 1.5-2 hours after a meal. The medication period was 4 weeks.
  Interventions: Drug: WPQW granule
- Control group (Placebo Comparator): Oral administration of WPQW granule simulant，which containing 5% WPQW granule，with warm water，2 sachets each time, 3 times a day, 1.5-2 hours after a meal. The medication period was 4 weeks.
  Interventions: Drug: WPQW granule simulant

INTERVENTIONS:
Drug: WPQW granule — WPQW granule, 2 sachets / time, 3 times / day.
  Arms: Experimental group
Drug: WPQW granule simulant — WPQW granule simulant, 2 sachets / time, 3 times / day.
  Arms: Control group

SUMMARY:
Non-erosive reflux disease（NERD）and Diarrhea-Predominant Irritable Bowel Syndrome（IBS-D）are both the common refractory gastrointestinal diseases. Patients, who suffered from overlapping symptoms of NERD and IBS-D, present more serious symptom manifestation, anxiety, and worse life quality than those with solely disease. There is lack of effective treatment for overlapping gastrointestinal symptoms. Traditional Chinese Medicine (TCM) syndrome differentiation and treatment has the advantages of overall regulation and individualized treatment, but lack of high-level evidence. The purpose of this study is to evaluate the efficacy and safety of WPQW granule for the treatment of NERD overlapping IBS-D.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a chronic relapsing acid-peptic disorder that is caused by the reflux of gastric or duodenum content. Non-erosive reflux disease（NERD）, which account for 70%, is the most common type of GERD in the Asian population. Diarrhea-Predominant Irritable Bowel Syndrome（IBS-D）is the mainly subtype of IBS, and the prevalence was found to be 46% in IBS. Both diseases aforementioned are common and frequent chronic diseases in the world, and the pathogenesis of which has not been fully defined. Current studies have shown that GERD can present in patients with IBS, vice versa. Up to 79% of patients with IBS co-exist with GERD-like symptoms, and 71% of patients with GERD co-exist with IBS-like symptoms. For those patients, they suffer from more serious symptom manifestation, anxiety, and worse life quality those with solely disease. The diagnosis and treatment of Functional gastrointestinal disorders (FGIDs) mostly based on the idea of segmental diagnosis and single-target therapy in modern medicine, and there is lack of effective treatment for overlapping gastrointestinal symptoms. The advantages of holistic diagnosis therapy and individualized treatment in Traditional Chinese Medicine（TCM）have attracted international attention, but there is still lack of high-level evidence-based medical evidence for the treatment of symptom overlap in FGIDs in TCM. In this study, we propose to conduct a multicenter, randomized, double-blind, placebo-controlled clinical study of WPQW granule for the treatment of NERD overlapping IBS-D to evaluate the efficacy and safety of WPQW granule with the aim of obtaining high-level evidence-based medical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with NERD and IBS-D simultaneously
2. Patients who present cardinal symptoms like reflux, heartburn, abdominal pain/bloating, diarrhea, etc
3. Patients diagnosed with syndrome of intermingled cold and heat of traditional Chinese medicine
4. Patients have informed consent and are willing to receive corresponding treatment

Exclusion Criteria:

1. Patients with hiatal hernia
2. Patients with upper gastrointestinal bleeding, peptic ulcer, gastrointestinal tumor, chronic atrophic gastritis with dysplasia
3. Patients with other serious organic diseases, such as acute cardiovascular disease, acute and chronic pancreatitis, cirrhosis, abnormal liver function (transaminases more than 1.5 times of normal value), abnormal thyroid function, diabetes mellitus with a history of more than 10 years, chronic renal insufficiency, hematologic disorders, and hematologic disorders, etc
4. Patients with neurological disease or psychiatric impairment like severe anxiety, depression requiring long-term drug treatment
5. Patients who cannot stop taking acid suppressants for a long time
6. Alcohol or drug dependency or abuse
7. Pregnant or lactating women
8. Patients who have a history of allergies to all the test drugs
9. Patients who are participating in other clinical trials or have participated in other clinical trials within 3 months
10. Patients who, in the opinion of the investigator, are not suitable to participate in clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change of visual analogue scale (VAS) score of symptoms of reflux and heartburn | baseline, 4 weeks during treatment period, 4 weeks during follow-up period
  During the medication period, the patients recorded the reflux and heartburn episodes (frequency and duration) within 24 hours per day on the symptom diary card, and VAS scores for reflux and heartburn symptoms was calculated as the mean score of each symptom in the past week. The episodes in the week before medication were used as the baseline, the mean score of any symptom decreased ≥50% from the baseline was recorded as response after weekly treatment, and the number of response weeks was considered effective if it was greater than 50% of the weeks of the whole treatment period.
Change of visual analogue scale (VAS) score of symptoms of abdominal pain and diarrhea | baseline, 4 weeks during treatment period, 4 weeks during follow-up period
  During the medication period, the patients recorded the of abdominal pain (pain severity and frequency) and diarrhea (stool consistency and frequency based on Bristol stool form scale) within 24 hours per day on the symptom diary card. VAS score was conducted for the most severe abdominal pain, and the mean score was calculated for each week, with the week of episodes prior to medication administration as the baseline. It was considered effective when the weekly mean score decrease of at least 30% from baseline and the days of at least once type 6 or type 7 stool Bristol stool form every week decrease of at least 30% from baseline, referring to the efficacy evaluation of the technical guidelines for clinical studies of Chinese medicine for IBS published in 2017.

SECONDARY OUTCOMES:
Change of traditional Chinese Medicine syndrome score | baseline, week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  The symptoms related to syndrome of intermingled cold and heat were scored. The cardinal symptom was scored 0, 2, 4, 6 and the secondary symptom scored 0, 1, 2, 3 respectively according to severity of each symptom. Total symptom score represented the syndrome score. Reduction in syndrome score represented Improvement.
Change of 36-item short-form (SF-36) score | baseline, week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Health status was evaluated by a 36-item short-form (SF-36) containing eight health concepts. If the score descends, it indicates that the patient's condition has improved.
Change of FGI-checklist score | baseline, week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  A 20-item FGI-checklist was used to evaluate comprehensive symptom severity of Functional Gastrointestinal Disorder (FGID), which covering esophageal, dyspeptic and bowel symptoms. If the score descends, it indicates that the patient's condition has improved.
Change of Hospital Anxiety and Depression Scale (HAD) score | baseline, week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Hospital Anxiety and Depression Scale (HAD) score was used to evaluate the efficacy of experimental drug. Reduction in total score represented Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Tang, M.D, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No